CLINICAL TRIAL: NCT04689464
Title: COVID19 and Psychological Health: a Cross Sectional Evaluation of the Risks of Anxiety and Depression Among Patients Diagnosed With Covid 19
Brief Title: COVID 19 and Psychological Health: a Cross Sectional Study to Evaluate Anxiety and Depression in Covid-19 Patients
Status: Completed | Type: Observational
Sponsor: Alhasan Mujtaba Al-Mudhaffer (Other)
Collaborators: University of Basrah (Other); Ministry of Health, Iraq (Network)
Responsible Party: Sponsor-Investigator, Alhasan Mujtaba Al-Mudhaffer, Clinical Pharmacy Specialist, AlFayhaa General Hospital
Organization: AlFayhaa General Hospital (Other)
Other Study IDs: 1120
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Anxiety; Depression
Keywords: COVID19; Anxiety; Depression
MeSH Terms: conditions — COVID-19; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild covid
- moderate covid
- severe covid

SUMMARY:
The covid-19 pandemic started to spread worldwide since December 2019. It promoted to an exaggerated psychological stress and anxiety in humans due to the intolerable symptoms higher than usual death of many infected patients. This study examines the corona related anxiety and if there is need for drug intervention to treat this anxiety.

To answer these questions, a survey made to the hospitalized patients including sex, age, educational level, Marital state, and a standardized questionnaires (GAD-7 and PHQ-9) which has been validated and shown to possess good psychometric qualities in studies of participants from multiple populations.

ELIGIBILITY:
Inclusion Criteria:

- patients with COVID19 willing to participate in the study

Exclusion Criteria:

* unwilling unable to read or interact with standardized questionnaire unconscious

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with covid19 diagnosed by their healthcare providers
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
depression | at the time of acute infection, average of 1 month
  Depression measured by Patient Health Questionnaire-9 (PHQ-9) scale. Scoring: 5-9 mild;10-14 moderate; 15-19 moderately severe; >20 severe. Minimum 0 maximum 27 points
anxiety | at the time of acute infection, average of 1 month
  Anxiety measured by General Anxiety Disorder-7 (GAD-7) scale. Scoring:5-9 mild; 10-14 moderate; >15 severe. Minimum 0, maximum 21 points

CONTACTS AND LOCATIONS:
Overall Officials: Zainab N Abdul-nabi, M.Sc., Study Director — University of Basrah; Hiba Dawood, M.Sc., Study Director — University of Basrah; Qussay N Almaliki, Ph.D., Study Director — AlFayhaa teaching hospital; Nadheera F Neamah, Study Director — University of Basrah; Dania Zydoon, Principal Investigator — Al-Sader teaching hospital; Zainab Mahdi, Principal Investigator — Al-Mawani general hospital
Locations (1):
- AlFayhaa Teaching hospital, Basra, Iraq

IPD SHARING:
Plan to Share IPD: Undecided